CLINICAL TRIAL: NCT01909193
Title: Cognitive Behavior Therapy vs. Attention Bias Modification Treatment for Social Anxiety
Brief Title: CBT vs. ABM vs. for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Associate Professor, Department of Psychology, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1624
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification (ABM) (Experimental): Attention training via 8 weekly repeated trials of a dot-probe task intended to direct attention away from threat stimuli.
  Interventions: Behavioral: Attention Bias Modification (ABM)
- Cognitive Behavior Therapy (Experimental): CBT will consist of 16-20 weekly individual treatment sessions aimed to reduce symptoms via cognitive and behavioral interventions
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Attention Bias Modification (ABM) — Attention training via 8 weekly repeated trials of a dot-probe task intended to direct attention away from threat stimuli.
  Arms: Attention Bias Modification (ABM)
Behavioral: Cognitive Behavior Therapy — CBT will consist of 16-20 weekly individual treatment sessions aimed to reduce symptoms via cognitive and behavioral interventions
  Arms: Cognitive Behavior Therapy

SUMMARY:
Adults with Social Anxiety Disorder will be pseudo randomly assigned to either an individual cognitive behavior therapy, attention bias modification treatment (allocation ratio - 1.5:1).

Outcome measures will be social anxiety symptoms and severity as measured by gold standard questionnaires as well as diagnosis of social anxiety disorder derived from structured clinical interviews based on Diagnostic and Statistical Manual (DSM) IV criteria.

The investigators expect to find significant reduction in social anxiety symptoms in all of the groups, with the cognitive behavior therapy group showing greater reduction in symptoms than the other groups. Mechanisms of change in all of the groups will be examined via measures of cognitive biases, affect, and other common and specific factors.

DETAILED DESCRIPTION:
120 Adults with Social Anxiety Disorder will be pseudo randomly assigned to either an individual cognitive behavior therapy (CBT), attention bias modification treatment (ABM)).

Outcome measures will be social anxiety symptoms and severity as measured by gold standard questionnaires as well as diagnosis of social anxiety disorder derived from structured clinical interviews based on DSM-IV criteria.

The investigators expect to find significant reduction in social anxiety symptoms in all of the groups, with the cognitive behavior therapy group showing greater reduction in symptoms than the other groups. Mechanisms of change in all of the groups will be examined via measures of cognitive biases, affect, and other common and specific factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Generalized Social Anxiety Disorder, LSAS>50
* If on medication, patients must be on a stable dose
* Hebrew language fluency

Exclusion Criteria:

* Primary Axis I or Axis II disorder other than SAD
* suicidal ideation
* Substance dependence within the past three months or current substance abuse
* Mental retardation or another pervasive developmental disability
* Current or past schizophrenia or psychosis, current bipolar disorder, or organic brain syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Liebovitz Social Anxiety Scale (LSAS) - diagnostic interview | Expected time frame of up to 32 weeks per participant. Participants will be assessed before and after the administration of the treatment, every 4 weeks during treatment and at 3 months follow-up
  LSAS is a 24-items clinician-administered scale developed for the assessment of fear and avoidance associated with social situations. The LSAS assesses a wide range of both social interaction and performance/observation situations, which are rated for degree of fear/anxiety and frequency of avoidance.

SECONDARY OUTCOMES:
Social Phobia Inventory (SPIN) - self-report questionnaire | Up to 32 weeks per participant. The SPIN will be administered before and after each treatment session and at 3 months follow-up
  The SPIN is a widely used 17-item self-report questionnaire that assesses fear, avoidance and physiological symptoms of social anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Huppert, PhD, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- The Hebrew University of Jerusalem, Jerusalem, Israel